CLINICAL TRIAL: NCT02527174
Title: A Phase I Study of Volasertib Combined With Standard Induction Chemotherapy for Previously Untreated Patients With Acute Myeloid Leukemia (VIAC)
Brief Title: A Study of Volasertib Plus Induction Chemotherapy for Acute Myeloid Leukemia
Acronym: VIAC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Volasertib no longer available
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Joseph Brandwein, Director, Division of Hematology, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230-37
Record Dates: First submitted 2015-07-06; First posted 2015-08-18 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — BI 6727; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study treatment arm (Experimental): Will receive volasertib combined with idarubicin plus cytarabine in a 3+7 schedule as induction chemotherapy. Volasertib dose will be given on day 4 in a dose escalation schedule over 3 dose levels (140 mg/m2, 170 mg/m2, 200 mg/m2) in successive cohorts.
  Non-hematologic toxicity will be determined using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 criteria for adverse events. Hematologic toxicity will be determined by days to absolute neutrophil count (ANC) and platelet recovery.
  Interventions: Drug: Volasertib; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Volasertib — Addition of single dose of volasertib intravenously (IV) on Day 4 of treatment protocol.
  Other Names: BI 6727
Drug: Idarubicin — Given IV daily on Days 1-3 of treatment protocol.
Drug: Cytarabine — Given IV daily as 24-hour continuous infusion on Day 1-7 of treatment protocol.
  Other Names: Ara-C

SUMMARY:
This is a Phase I clinical trial to determine the maximum tolerated dose (MTD) of the polo-like kinase-1 inhibitor volasertib which can be safely combined with idarubicin plus cytarabine induction chemotherapy for previously untreated patients with acute myeloid leukemia. (AML).

DETAILED DESCRIPTION:
Main inclusion criteria:

1. AML, any subtype except acute promyelocytic leukemia (APL)
2. At least one of the following features:

   i. Age 18-75 with adverse risk cytogenetics ii. Age 18-75 with antecedent myelodysplastic syndrome (MDS) or myeloproliferative disorder (MPD), or therapy-related AML iii. Age 60-75, regardless of risk category
3. No prior therapy for AML other than hydroxyurea
4. Judged by treating physician to be medically fit for induction chemotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2
6. Normal left ventricular ejection fraction

Subjects will receive induction chemotherapy consisting of idarubicin 12 mg/m2 on Days 1-3 plus cytarabine 200 mg/m2 (age 18-59) or 100 mg/m2 (age 60-75) as a continuous IV infusion x 7 days. Volasertib will be administered on day 4 in a dose-escalation schedule, using a standard 3+3 dose escalation design, over 3 dose levels. Once the MTD has been determined, an additional dose expansion cohort will be accrued.

ELIGIBILITY:
Inclusion Criteria:

1. AML, any World Health Organization (WHO) subtype except APL, either de novo or secondary; extramedullary AML (i.e. granulocytic sarcoma) is permitted.
2. At least one of the following features:

   * Age 18-75 with adverse risk cytogenetics, including:

     * Complete or partial deletion of chromosome 5 or 7
     * Complex karyotype, defined as > 3 abnormalities, excluding t(15;17). t(8;21) or inv(16) or variant
     * 11q23 abnormality
     * Inv(3)(q21;q26) or variant
     * t(6;9)
     * abn(17p)
   * Age 18-75 with secondary AML, defined as arising from an antecedent myelodysplastic syndrome (MDS) or myeloproliferative disorder (MPD), or therapy-related AML
   * Age 60-75, regardless of risk category
3. No prior therapy for AML other than hydroxyurea (allowed for up to 28 days). Prior therapy for MDS, MPD or other malignancy is allowed.
4. Judged by treating physician to be medically fit for induction chemotherapy
5. ECOG performance status score 0-2.
6. Left ventricular ejection fraction (LVEF) within normal limits, by myocardial multigated scan (MUGA) or echocardiogram.
7. Signed and dated written informed consent prior to admission

Exclusion Criteria:

1. Prior anthracycline exposure equivalent to > 300 mg/m2 doxorubicin.
2. Prior chemotherapy or radiotherapy within previous four weeks except for hydroxyurea.
3. Prior treatment with volasertib or any other Polo-like kinase inhibitor
4. Known hypersensitivity to the trial drug
5. Serum creatinine > 1.5 times (1.5x) upper limit of normal (ULN) or creatinine clearance (CLcr) < 30 ml/min (estimated creatinine clearance by the Cockcroft-Gault (C-G) equation
6. Serum bilirubin > 1.5x ULN, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x ULN
7. Persistence of clinically relevant therapy related toxicity from previous anti-cancer therapy
8. Active central nervous system leukemia (no lumbar puncture required; clinical judgement is sufficient)
9. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
10. Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure (> New York Heart Association-II), serious cardiac arrhythmia, pericardial effusion)
11. QTcF prolongation > 470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).The QTcF will be calculated as the mean of the 3 ECGs taken at screening.
12. Other concurrent malignancy requiring active therapy (except hormonal therapy for prostate or breast cancer).
13. Severe uncontrolled infection. Controlled infection on antibiotics is permitted.
14. Active or chronic hepatitis C and/or B infection
15. Known HIV infection
16. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
17. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least six months after end of active therapy on study.
18. Pregnancy or breast feeding, female patients must have a negative pregnancy test prior to commencing study treatment.
19. Psychological, familial or sociological factors potentially hampering compliance with the study protocol and follow-up schedule
20. Known or suspected active alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile | Participants will be followed for duration of induction cycle (expected time 28-35 days) for toxicity.
  Non-hematologic toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Hematologic toxicities will be assessed by determining number of days to neutrophil (ANC) recovery to >0.5 x10(9)/L or platelet recovery to >20 x10(9)/L.
Dose-limiting toxicity (DLT) | Participants will be followed for duration of induction cycle (expected time 28-35 days) for DLT assessment.
  DLT is defined as grade 3-4 non-hematologic toxicity (except grade 3 nausea, vomiting, mucositis or creatinine elevation due to tumor lysis syndrome, and grade 3-4 neutropenic infections and electrolyte abnormalities) using CTCAE version 4.0.Hematologic DLT is defined as ANC recovery to >0.5 x10(9)/L or platelet recovery to >20 x10(9)/L of > 42 days.
Maximum tolerated dose (MTD) | Determined after completion of dose-escalation phase of study, which will take approx. 12-15 months.
  MTD is defined as maximum dose of volasertib associated with < 2/6 DLTs at a given dose level.

SECONDARY OUTCOMES:
Complete response rate of regimen | Responses will be determined at hematologic recovery (Day 28 or greater, up to Day 60).
  Complete response (CR) defined as <5% marrow blasts with ANC > 1.0 x10(9)/L and platelets >100 x 10(9)/L, with no extramedullary disease. CRi defined as same, but ANC <1.0 and/or platelets <100.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Brandwein, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available to Boehringer-Ingelheim.